CLINICAL TRIAL: NCT05246306
Title: Comparison of Aerobic Capacity and Physical Fitness Level of Adolescents With Polycystic Ovary Syndrome and Healthy Peers
Brief Title: Aerobic Capacity and Physical Fitness Level of Adolescents With PCOS
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Dr. Sami Ulus Children's Hospital (Other)
Responsible Party: Principal Investigator, Ebru Calik Kutukcu, Associate Professor, Hacettepe University
Other Study IDs: GO 21/947
Record Dates: First submitted 2022-01-21; First posted 2022-02-18 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Polycystic Ovary Syndrome
Keywords: aerobic capacity; physical fitness
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy group: Healthy adolescents aged 14-24 who have not been diagnosed with any chronic disease
- Patient with PCOS group: Adolescents between the ages of 14-24 diagnosed with Polycystic Ovary Syndrome according to the Rotherdam criteria.

SUMMARY:
Polycystic Ovary Syndrome (PCOS) is associated with hyperandrogenism, hyperinsulinemia and insulin resistance starting in the perimenarchal period. Insulin resistance also increases the risk of developing glucose intolerance, type 2 diabetes, hypertension, dyslipidemia and cardiovascular disorders. Studies on adult women with PCOS show that their aerobic capacity is affected. Therefore, in this study; it was aimed to compare the physical and cardiovascular fitness levels of adolescent PCOS patients with healthy adolescents.

DETAILED DESCRIPTION:
Polycystic Ovary Syndrome (PCOS) is associated with hyperandrogenism, hyperinsulinemia and insulin resistance starting in the perimenarchal period. Insulin resistance also increases the risk of developing glucose intolerance, type 2 diabetes, hypertension, dyslipidemia and cardiovascular disorders. Studies on adult women with PCOS show that their aerobic capacity is affected. Therefore, in this study; it was aimed to compare the physical and cardiovascular fitness levels of adolescent PCOS patients with healthy adolescents.Total fat and muscle ratios will be measured with the bioelectrical impedance test (BIA) instrument for body composition evaluation of individuals in both groups. Body mass index (BMI), waist/hip and waist/height ratios will be recorded. The level of cardiovascular fitness will be evaluated with the PACER test, which is among the Fitness Gram Test Protocol. For physical fitness level, muscular strength parameter will be evaluated with hand dynamometer and knee extensor muscle strength, and muscular endurance parameter will be evaluated with sit-up and push-up tests. Participants' physical activities will be evaluated with the Adolescent Physical Activity Questionnaire (PAQ-A).The quality of life of individuals with PCOS will be evaluated with the Polycystic Ovary Syndrome Quality of Life-50 Scale.

ELIGIBILITY:
Inclusion Criteria of patients :

* Being between the ages of 14-24,
* Collecting Polycystic Syndrome according to Rotherdam,
* Not having had Covid-19.

Exclusion Criteria of the patients :

* Not to be between the ages of 14-24,
* Not showing the symptoms of Polycystic Ovary Syndrome (PCOS),
* Having had Covid-19,
* Having a chronic disease diagnosed other than PCOS,
* Having cognitive impairment that will affect their cooperation with tests.

Healthy group inclusion criteria

* Being a female adolescent between the ages of 14-24,
* Not having been diagnosed with any chronic disease,
* Adolescents with regular menstrual cycles,
* Not taking any medication known to affect hormone, lipid and carbohydrate metabolism,
* Not having clinical signs of hyperandrogenism,
* Not having had Covid-19.

Healthy group exclusion criteria

* Not to be between the ages of 14-24,
* Having a chronic disease,
* Having had Covid-19,
* Having cognitive impairment that will affect their cooperation with tests.

Ages: 14 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy group: Being in the adolescent group, not having any chronic disease and being willing to participate in the study.
  Patient group: Being in the adolescent group, being diagnosed with polycystic ovary syndrome and being willing to participate in the study
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Aerobic Exercise Capacity | 1 day
  PACER running test, which is included in the fitnessgram test protocol, will be used to evaluate aerobic capacity.
Physical Fitness | 1 day
  The Fitnessgram Test Protocol will be used for physical fitness assessment.

SECONDARY OUTCOMES:
Peripheral Muscle Strength | 1 day
  With the Lafayette Manual Muscle Test System Model01165, knee extensor muscle strength will be measured in individuals in sitting position and knee extension. 3 repetitions will be applied for the right and left sides and the results will be recorded in kilograms.
Physical Activity Level | 1 day
  Adolescent Physical Activity Questionnaire (PAQ-A) will be administered to both groups. This questionnaire is designed to assess physical activity in the last 7 days. It consists of 8 questions in which the answers given are scored between 1 and 5, and 9 questions questioning the existence of a situation that prevents physical activity in the last week.
Life quality | 1 day
  The quality of life of individuals with Polycystic Ovary Syndrome will be evaluated with the Polycystic Ovary Syndrome Quality of Life-50 Scale. This scale consists of six parameters including psychosocial and status, fertility, sexual function, obesity and menstrual irregularity, hair growth and coping with the disease, and includes 50 questions. When calculating the total score and sub-dimension scores of the scale, it is scored as 5 never, rarely 4, sometimes 3, often 4, always 1.
Body composition analysis | 1 day
  Body fat percentage (%), body muscle percentage (%), body water percentage (%), body fat weight (kg), body muscle weight (kg) will be recorded according to Bioelectrical Impedance Analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Calik Kutukcu, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No